CLINICAL TRIAL: NCT03114202
Title: Effects of Intensive Nutritional Counseling on Nutritional Status and Quality of Life of Patients With Head and Neck Cancer Undergoing Radiation Therapy
Brief Title: Effects of Nutritional Counseling on Nutritional Status and Quality of Life of Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.954.066
Record Dates: First submitted 2017-03-23; First posted 2017-04-14 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intensive nutritional counseling: once they are admitted to the study and once a week during radiotherapy
  Interventions: Other: intensive nutritional counseling
- Control group (Other): Standard care: when there is demand, usually 1 to 2 times during radiotherapy
  Interventions: Other: Standard care

INTERVENTIONS:
Other: intensive nutritional counseling — Individualised nutrition intervention in the form of regular and intensive nutrition counselling by a dietitian, following a predetermined standard nutrition protocol, the Medical Nutrition Therapy (Cancer/Radiation Oncology) protocol of the American Dietetic Association (ADA) every week during radiotherapy. Individually tailored sample meal plans, recipe suggestions and hints to minimise the side effects of the tumour and therapy will be provided.
  Arms: Intervention group
Other: Standard care — Nutritional counseling / education performed by hospital nurses and nutritional care performed by the hospital nutritionist.
  Arms: Control group

SUMMARY:
This study investigates the effects of nutritional counseling versus standard nutritional care on nutritional status and quality of life in patients with head and neck cancer submitted to radiotherapy.Half participants will receive intensive nutritional counseling while the other half will receive standard care.

DETAILED DESCRIPTION:
Considering that head and neck cancer patients usually present reduced food intake with consequent involuntary weight loss and significant worsening of quality of life, this study investigates the effects of nutritional counseling versus standard nutritional care on nutritional status and quality of life in patients with head and neck cancer submitted to radiotherapy.

Half participants (45) will receive intensive nutritional counseling, that is, once they are admitted to the study and once a week during radiotherapy, following the protocol of nutritional care to cancer patients in radiotherapy proposed by the American Dietetic Association (ADA).

The other half (45) will receive standard care, that is, nutritional counseling / education performed by hospital nurses and nutritional care performed by the hospital nutritionist (when there is a demand, usually 1 to 2 times during oncologic treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer (oral cavity, oropharynx, hypopharynx and larynx); both sexes; aged 18 years and over, submitted to radiotherapy after chemotherapy or radiotherapy as a first-choice treatment or as adjuvant treatment (post-surgical).

Exclusion Criteria:

* Patients using parenteral nutrition; without cognitive ability to understand the concepts of the questionnaires; in palliative radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-08-06 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline and 12 weeks
  Defined as mean weight change
Change in nutritional status | Baseline and 12 weeks
  Defined as mean body mass index change
Change in quality of life | Baseline and 12 weeks
  Self reported quality of life assessed using two questionnaires - Functional Assessment of Cancer Therapy - Head and Neck (FACT-H & N) and European Organization for Research and Treatment of Cancer - Quality of life questionnaire - Head and Neck (EORTC-QLQ-H & N35).

SECONDARY OUTCOMES:
Change in patient generated subjective global assessment | Baseline and 12 weeks
  Self reported nutritional assessment by the Scored Patient-Generated Subjective Global Assessment (PG-SGA)
Energy and protein intake | Baseline and 12 weeks
  Mean changes in energy and protein intake, assessed by the 24 hour recording
Fat free mass | Baseline and 12 weeks
  Mean changes in fat free mass, assessed by foot-to-foot bioimpedance
Occurrence of complications due to radiotherapy | 12 weeks
  Number of patients with complications due to radiotherapy, assessed from medical record
Occurrence of unplanned hospitalization | 12 weeks
  Number of patients with unplanned hospitalization, assessed from medical record
Occurrence of interruption or delay in treatment. | 12 weeks
  Number of patients with interruption or delay in treatment, assessed from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Jose Eluf Neto, Principal Investigator — São Paulo University; Andre Carvalho, Study Chair — Hospital de Cancer de Barretos - Fundação PIO XII; Sheilla Faria, Study Chair — São Paulo University
Locations (2):
- Brazil (2):
  - Centro de Oncologia da Santa Casa Nossa Senhora do Perpétuo Socorro, Alfenas, Minas Gerais
  - Fundação Hospitalar do Município de Varginha - Hospital Bom Pastor, Varginha, Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided